CLINICAL TRIAL: NCT01228760
Title: A Phase 1, Open-label, Multi-center, Dose Escalation Study of the Safety and Pharmacokinetics of ASG-5ME Monotherapy in Subjects With Castration-Resistant Prostate Cancer (CRPC)
Brief Title: A Study to Determine the Maximum Tolerated Dose of ASG-5ME in Subjects With Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASG-5ME-10-1
Record Dates: First submitted 2010-10-21; First posted 2010-10-26 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Neoplasms
Keywords: Castration-Resistant Prostate Cancer; ASG-5ME; Pharmacokinetics of ASG-5ME
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ASG-5ME

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Dose level 1 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 2 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 3 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 4 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 5 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 5A (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 6 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 7 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 8 (Experimental)
  Interventions: Drug: ASG-5ME
- Dose level 9 (Experimental)
  Interventions: Drug: ASG-5ME
- Chemotherapy-naïve subjects (Experimental)
  Interventions: Drug: ASG-5ME
- Chemotherapy exposed subjects (Experimental)
  Interventions: Drug: ASG-5ME

INTERVENTIONS:
Drug: ASG-5ME — IV

SUMMARY:
The purpose of this dose escalation study is to determine the Maximum Tolerated Dose (MTD) and the recommended Phase 2 dose of ASG-5ME in subjects with castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
The study has two components. The first aims to establish a safe dose of ASG-5ME. Once identified, the safety and preliminary estimate of antitumor activity of ASG-5ME will be tested in additional subjects with castration-resistant prostate cancer (CRPC) who are either chemotherapy naïve or chemotherapy exposed in expanded cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically-confirmed castration-resistant prostate cancer and meets at least 1 of the following criteria:

  * subject's disease has progressed on or after available standard therapy -OR-
  * there is no effective standard therapy available for treating the subject's disease -OR-
  * subject or his disease is not suitable for standard therapy -OR-
  * subject chooses to defer or decline standard therapy (subject is adequately informed of the availability of clinically meaningful therapy and chooses instead to partake in this research using a product with no documented clinical activity)
* Testosterone ≤ 50 ng/dL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of > 6 months as evaluated and documented by the investigator
* Hematologic function, as follows (no red blood cell (RBC) or platelet transfusions are allowed within 4 weeks of the first dose of ASG-5ME):

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL
* Renal function, as follows: creatinine ≤ 1.5 x upper limit of normal (ULN), or creatinine clearance of > 60 mL/min if serum creatinine is > 2.0 mg/dL
* Total bilirubin < 1. 5 x ULN
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT)≤ 1.5 x ULN
* International Normalized Ratio (INR) < 1.3 (or < 3.0 if on therapeutic anticoagulation)
* Serum calcium ≤ ULN
* Subjects must be taking and agree to remain on a stable dose of luteinizing hormone-releasing hormone (LHRH) agonist therapy or gonadotropin-releasing hormone (GnRH) antagonist for the duration of the trial if not surgically castrated
* Additional Inclusion criteria for Chemotherapy Naïve Cohort: No prior systemic cytotoxic chemotherapies
* Additional Inclusion criteria for Chemotherapy Exposed Cohort:

  * Documented disease progression during or after docetaxel treatment or intolerability to docetaxel treatment
  * No additional prior chemotherapy for CRPC is allowed

Exclusion Criteria:

* History of central nervous system metastasis, including incompletely treated epidural disease
* History of other primary malignancy (including premalignant myeloid malignancy e.g. myelodysplastic syndrome), unless:

  * Curatively resected non-melanomatous skin cancer
  * Other malignancy curatively treated with no known active disease present and no treatment administered for the last 3 years
* Active angina or Class III or IV Congestive Heart Failure (CHF) (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 12 months of study enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrhythmias not controlled by outsubject medication
* The following treatments are not allowed within 4 weeks of enrollment: cytotoxic chemotherapy, radiation therapy or the dietary supplement PC-SPES
* Use of prednisone (or equivalent corticosteroids) > 20 mg/day are not allowed. Doses < 20 mg/day are allowed only if they have been at the same dose for > 4 weeks
* Use of anti-androgen therapy (ie, flutamide, bicalutamide and nilutamide) within 6 weeks of study enrollment; non-responders to second-line anti-androgen therapy do not require the 6 week withdrawal period
* Monoclonal antibody therapy within 3 months of enrollment with the exception of denosumab (prior or concurrent use of denosumab is allowed)
* Peripheral neuropathy of ≥ grade 2 as defined by the CTCAE criteria version 4.0
* Major surgery (that requires general anesthesia) within 4 weeks of study enrollment
* Active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, or antiviral agent) within 72 hours of screening
* Use of any investigational drug (including marketed drugs not approved for this indication) within 30 days prior to enrollment
* History of thromboembolic events and bleeding disorders ≤ 3 months (e.g., deep vein thrombosis (DVT) or pulmonary embolism (PE))
* Known positive test for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B surface antigen

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Safety assessed by recording of adverse events, laboratory assessments and vital signs | For 12 weeks during treatment period and up to 4 weeks follow up
Pharmacokinetics assessment of ASG-5ME blood levels through analysis of blood samples | Up to day 15 for cycle 1 and cycle 4 and pre-dose for cycles 2 and 3; every 3 weeks during the second 12 weeks of treatment; and if subject continues on study drug, every 12 weeks thereafter

SECONDARY OUTCOMES:
Incidence of anti-ASG-5ME antibody formation | Baseline; up to day 64 during the first 12 weeks; and if subject continues on study drug, every 3 weeks during the second 12 weeks of treatment and every 12 weeks thereafter
Incidence of tumor response (complete or partial response) | Baseline and every 12 weeks while on study drug
Changes in prostate-specific antigen (PSA) levels | Baseline; up to day 64 during the first 12 weeks; and if the subject continues on study drug, every 3 weeks thereafter
Changes in bone scans | Baseline and every 12 weeks while on study drug
Changes in circulating tumor cells | Baseline; up to day 64 during the first 12 weeks; and if the subject continues on study drug, every 3 weeks during the second 12 weeks of treatment and every 12 weeks thereafter
Changes in cytokeratin-18 levels | Up to day 79 and 4 weeks after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Agensys, Inc.
Locations (4):
- United States (4):
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - The Karmanos Cancer Institute, Detriot, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Wisconsin Madison, Carbone Cancer Center, Madison, Wisconsin